CLINICAL TRIAL: NCT03362593
Title: A Phase 1 Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of MEDI7219 in Healthy Subjects, Including Assessment of the Impact of Changes to the Oral Formulation and Determination of Intravenous Pharmacokinetics
Brief Title: A 6-Part Study In Healthy Volunteers To Evaluate Safety, Tolerability and Uptake Of MEDI7219 in the Body When Given as Single and Multiple Doses
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The program is canceled due to company strategic reasons.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D8170C00001
Record Dates: First submitted 2017-11-22; First posted 2017-12-05 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — MEDI7219; Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MEDI7219 (Experimental): Experimental Drug
  Interventions: Drug: MEDI7219
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Formulation without Active Drug (Placebo Comparator): Formulation without Active Drug
  Interventions: Drug: Formulation without Active Drug

INTERVENTIONS:
Drug: MEDI7219 — Experimental Drug
  Arms: MEDI7219
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Formulation without Active Drug — Formulation without Active Drug
  Arms: Formulation without Active Drug

SUMMARY:
This is a 6-part study to evaluate the safety, tolerability, and PK of MEDI7219 in healthy subjects. Parts A, B, C & E are the single-dose parts of the study. Parts D & F are the multiple ascending dose (MAD) parts of the study. The starting dose and formulation for Parts D & F will be selected from data emerging from Parts A, B and E. Enrollment of approximately 198 subjects is anticipated.

DETAILED DESCRIPTION:
MEDI7219 is being developed for the potential treatment of type 2 diabetes. The study is a first in human, single and multiple ascending dose study that will try to identify the safety, tolerability and pharmacokinetics (how the drug moves through the body) of MEDI7219. The study will also look at the impact of changes to the formulation as well as differences related to the route of administration. The study will consist of 6 parts involving approximately 198 healthy male and female subjects (and up to 146 additional subjects). In Part A, 6 cohorts of 10 subjects each (with an optional 2 cohorts) will be randomized to receive MEDI7219 or one of two placebos. Each cohort will receive a different formulation of the study drug. In part B, a single cohort of 16 subjects (with an optional second cohort) will receive a different formulation of MEDI7219 per period in up to 5 periods. In Part C, up to 12 subjects will be dosed with MEDI7219. In Part D, one cohort of 30 subjects (with an optional second cohort) will be randomized to receive MEDI7219 or placebo. Subjects will start on a dose based on data from previous parts and will receive ascending doses for 35 days. In Part E, 2 cohorts of 6 subjects each (with an optional third & fourth cohort of 12 subjects each) will receive a different formulation of MEDI7219 per period. Part E, cohort 5 12 subjects each period (2 periods) has been added to assess 2 different formulations In Part F, two cohorts of 16 subjects each will be randomized to receive MEDI7219 or placebo. Subjects will start on a dose based on data from previous parts and will receive ascending doses for 35 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers age 18-55 years
* BMI 18-32 kg/m2
* Females not of childbearing potential
* Able and willing to adhere to the protocol
* Must provide written informed consent

Exclusion Criteria:

* Any concurrent condition that in the opinion of the investigator would interfere with the evaluation of the investigational product
* Abnormal lab values, physical exam, vital signs
* Positive drug or alcohol screen.
* Current enrollment in another clinical study or enrollment within the past 3 months
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks prior to dosing
* Abnormal ECG
* Positive Hepatitis B, Hepatitis C or HIV test
* Positive Drug or Alcohol screen
* Current smokers or those who have smoked within the last 12 months
* Recent plasma or blood donation
* Evidence of current SARS-CoV-2 infection (Part E Cohort 5 and Part F Cohort 2 only)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 186 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events as a measure of safety and tolerability of MEDI7219 | Baseline to last follow up visit (Parts A and C - Day 28) (Part D & F Day 63) and (Parts B and E 28 days post last dose)
  Treatment emergent adverse events (TEAEs) and serious adverse events (TESAEs)

SECONDARY OUTCOMES:
Pharmacokinetics of MEDI7219: Cmax | Pre-dose to 144 hours post-dose (Parts A, B, C and Part E cohorts 1 & 2 only); Pre-dose to 168 hours post-dose (Part E optional cohorts only); Parts D & F pre-dose to Day 63/EOS visit
  PK parameters will be calculated from the plasma concentration versus time data for Cmax (maximum observed concentration)
Pharmacokinetics of MEDI7219: Tmax | Pre-dose to 144 hours post-dose (Parts A, B, C and Part E cohorts 1 & 2 only); Pre-dose to 168 hours post-dose (Part E optional cohorts only); Parts D & F pre-dose to Day 63/EOS visit, Parts F cohort 2 ONLY: Pre-dose and 8 hours post-dose
  PK parameters will be calculated from the plasma concentration versus time data for Tmax (time to maximum observed concentration)
Pharmacokinetics of MEDI7219: t1/2 | Pre-dose to 144 hours post-dose (Parts A, B, C and Part E cohorts 1 & 2 only); Pre-dose to 168 hours post-dose (Part E optional cohorts only); Parts D & F pre-dose to Day 63/EOS visit
  PK parameters will be calculated from the plasma concentration versus time data for T1/2 (terminal half-life)
Pharmacokinetics of MEDI7219: AUC (0-inf) | Pre-dose to 144 hours post-dose (Parts A, B, C and Part E cohorts 1 & 2 only); Pre-dose to 168 hours post-dose (Part E optional cohorts only); Parts D & F pre-dose to Day 63/EOS visit
  PK parameters will be calculated from the plasma concentration versus time data for AUC (0-inf) [area under the curve (AUC) extrapolated to infinity]
Pharmacokinetics of MEDI7219: AUC(0-last) | Pre-dose to 144 hours post-dose (Parts A, B, C and Part E cohorts 1 & 2 only); Pre-dose to 168 hours post-dose (Part E optional cohorts only); Parts D & F pre-dose to Day 63/EOS visit
  PK parameters will be calculated from the plasma concentration versus time data for AUC (0-last) [area under the curve (AUC) from time 0 to last measurable concentration]
Pharmacokinetics of MEDI7219: AUC(0-24h) | Pre-dose to 144 hours post-dose (Parts A, B, C and Part E cohorts 1 & 2 only); Pre-dose to 168 hours post-dose (Part E optional cohorts only); Parts D & F pre-dose to Day 63/EOS visit
  PK parameters will be calculated from the plasma concentration versus time data for (AUC 0-24) [area under the curve (AUC) from time 0 to 24 hours post dose]
Pharmacokinetics of MEDI7219: AUC (%extrap) | Pre-dose to 144 hours post-dose (Parts A, B, C and Part E cohorts 1 & 2 only); Pre-dose to 168 hours post-dose (Part E optional cohorts only)
  PK parameters will be calculated from the plasma concentration versus time data for AUC%extrapolated [The percentage of AUC(0-inf) accounted for by extrapolation]
Pharmacokinetics of MEDI7219: Lambda-z | Pre-dose to 144 hours post-dose (Parts A, B, C and Part E cohorts 1 & 2 only); Pre-dose to 168 hours post-dose (Part E optional cohorts only)
  PK parameters will be calculated from the plasma concentration versus time data for Lambda-z [Slope of the regression line passing through the apparent elimination phase in a concentration vs time plot]
Pharmacokinetics of MEDI7219: CL/F | Pre-dose to 144 hours post-dose (Parts A, B and Part E cohorts 1 & 2 only); Pre-dose to 168 hours post-dose (Part E optional cohorts only)
  PK parameters will be calculated from the plasma concentration for CL/F (apparent clearance)
Pharmacokinetics of MEDI7219: Vz/F | Pre-dose to 144 hours post-dose (Parts A, B and Part E cohorts 1 & 2 only); Pre-dose to 168 hours post-dose (Part E optional cohorts only); Pre-dose to Day 63/EOS visit (Parts D & F)
  PK parameters will be calculated from the plasma concentration for Vz/F (volume of distribution)
Pharmacokinetics of MEDI7219: Frel | Pre-dose to 144 hours post-dose (Parts B and Part E cohorts 1 & 2 only); Pre-dose to 168 hours post-dose (Part E optional cohorts only)
  PK parameters will be calculated from the plasma concentration for Frel (relative bioavailability)
Pharmacokinetics of MEDI7219: Vd | Pre-dose to 144 hours (Part C)
  PK parameters will be calculated from the plasma concentration for Vd (volume of distribution)
Pharmacokinetics of MEDI7219: F | Pre-dose to 144 hours (Part C )
  PK parameters will be calculated from the plasma concentration for F (absolute bioavailability)
Pharmacokinetics of MEDI7219: AUC (0-tau) | Pre-dose to Day 63/EOS visit (Parts D & F)
  PK parameters will be calculated from the plasma concentration versus time data for AUC (0-tau) [area under the curve (AUC) for a dosing interval]
Immunogenicity | Day -1 to Day 28/EOS Visit (Parts A and C); Day -1 to Day 63/EOS Visit (Parts D & F); Day -1 to 28 days post last dose of final period/EOS Visit (Parts B and E)
  Presence of Anti-drug antibody to MEDI7219
Pharmacokinetics of Formulation Component: Cmax | Predose to 8 hours post dose Day 1 (Parts A, B and E); Pre-dose to 8 hours post dose on Days 1, 7, 8, 14, 15, 21, 22, 28, 29 and 35 (Part D and F Cohort 1); Pre-dose to 24 hours post dose on Days 1, 14, 28 and 35 (Part F Cohort 2, respectively)
  PK parameters will be calculated from the plasma concentration versus time data for Cmax (maximum observed concentration)
Pharmacokinetics of Formulation Component: Tmax | Predose to 8 hours post dose Day 1 (Parts A, B and E); Pre-dose to 8 hours post dose on Days 1, 7, 8, 14, 15, 21, 22, 28, 29 and 35 (Part D and F Cohort 1); Pre-dose to 24 hours post dose on Days 1, 14, 28 and 35 (Part F Cohort 2, respectively)
  PK parameters will be calculated from the plasma concentration versus time data for Tmax (time to maximum observed concentration)
Pharmacokinetics of Formulation Component: T(1/2) | Predose to 8 hours post dose Day 1 (Parts A, B and E); Pre-dose to 8 hours post dose on Days 1, 7, 8, 14, 15, 21, 22, 28, 29 and 35 (Part D and F Cohort 1); Pre-dose to 24 hours post dose on Days 1, 14, 28 and 35 (Part F Cohort 2, respectively)
  PK parameters will be calculated from the plasma concentration versus time data for T1/2 (terminal half-life)
Pharmacokinetics of Formulation Component: AUC (0-inf) | Predose to 8 hours post dose Day 1 (Parts A, B and E); Pre-dose to 8 hours post dose on Days 1, 7, 8, 14, 15, 21, 22, 28, 29 and 35 (Part D and F Cohort 1); Pre-dose to 24 hours post dose on Days 1, 14, 28 and 35 (Part F Cohort 2, respectively)
  PK parameters will be calculated from the plasma concentration versus time data for AUC (0-inf) [area under the curve (AUC) extrapolated to infinity]
Pharmacokinetics of Formulation Component: AUC (0-last) | Predose to 8 hours post dose Day 1 (Parts A, B and E); Pre-dose to 8 hours post dose on Days 1, 7, 8, 14, 15, 21, 22, 28, 29 and 35 (Part D and F Cohort 1); Pre-dose to 24 hours post dose on Days 1, 14, 28 and 35 (Part F Cohort 2, respectively)
  PK parameters will be calculated from the plasma concentration versus time data for AUC (0-last) [area under the curve (AUC) from time 0 to last measurable concentration]
Pharmacokinetics of Formulation Component: AUC (0-8h) | Predose to 8 hours post dose Day 1 (Parts A, B and E); Pre-dose to 8 hours post dose on Days 1, 7, 8, 14, 15, 21, 22, 28, 29 and 35 (Part D and F Cohort 1); Pre-dose to 24 hours post dose on Days 1, 14, 28 and 35 (Part F Cohort 2, respectively)
  PK parameters will be calculated from the plasma concentration versus time data for (AUC 0-24) [area under the curve (AUC) from time 0 to 8 hours post dose]
Pharmacokinetics of MEDI7219: CL | Pre-dose to 144 hours post-dose (Part C)
  PK parameters will be calculated from the plasma concentration from CL (apparent clearance)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ standards.
Supporting Information: ICF
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Mou S, Hummer BT, Yuan J, Huang Y, Liang M, Faggioni R, Roskos LK, Rosenbaum AI. Investigations of Enteric-Coated Tablet Propyl Gallate-Induced Nephrotoxicity in Beagles as well as Human and Dog Renal Proximal Tubule Epithelial Cells. ACS Pharmacol Transl Sci. 2025 Apr 4;8(5):1282-1291. doi: 10.1021/acsptsci.4c00563. eCollection 2025 May 9. PMID 40370985